CLINICAL TRIAL: NCT07258446
Title: PRAME (Preferentially Expressed Antigen in Melanoma) Immunohistochemistry Guided Slow-Mohs Micrographic Surgery of Malignant Melanoma: A Pragmatic Clinical Trial
Brief Title: PRAME Immunohistochemistry-Guided Slow Mohs Micrographic Surgery for the Treatment of Stage 0 to IIc Cutaneous Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC324; NCI-2025-08321 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC324 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Clinical Stage 0 Cutaneous Melanoma AJCC v8; Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — Immunohistochemistry; Mohs Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (PRAME IHC-guided SMMS) (Experimental): Patients undergo standard slow Mohs micrographic surgery with the addition of PRAME IHC analysis per the discretion of the surgeon on study.
  Interventions: Diagnostic Test: Immunohistochemistry Staining Method; Procedure: Mohs Surgery

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry Staining Method — Undergo Preferentially Expressed Antigen in Melanoma (PRAME) IHC analysis
  Other Names: Cell/Tissue, Immunohistochemistry; IHC; Immunohistochemistry; Immunohistochemistry (IHC); PRAME; Preferentially Expressed Antigen in Melanoma
Procedure: Mohs Surgery — Undergo slow Mohs micrographic surgery
  Other Names: Mohs Micrographic Surgery

SUMMARY:
This clinical trial tests the addition of preferentially expressed antigen in melanoma (PRAME) immunohistochemical (IHC) staining to standard slow Mohs micrographic surgery (SMMS) for guiding tissue removal in patients with stage 0 to IIc cutaneous melanoma. SMMS is a method of skin cancer removal involving repeated tissue removal and examination under a microscope to ensure the tumor is removed as much as possible while sparing healthy tissue. In SMMS, tissue sections are evaluated to determine whether additional tissue removal is needed. The standard method for evaluating the tissue is by using a specific stain called hematoxylin and eosin (H&E) stains. PRAME is a cancer antigen that is being investigated as a diagnostic marker in certain types of cancer. Adding PRAME IHC analysis to standard SMMS staining methods may improve the accuracy for determining whether additional tissue removal is necessary for patients undergoing SMMS for stage 0 to IIc cutaneous melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the efficacy of PRAME IHC-guided slow Mohs micrographic surgery to routine slow Mohs micrographic surgical practices in patients with melanoma.

SECONDARY OBJECTIVE:

I. To further evaluate the efficacy of PRAME IHC-guided slow Mohs micrographic surgical practices in patients with melanoma.

OUTLINE:

Patients undergo standard slow Mohs micrographic surgery with the addition of PRAME IHC analysis per the discretion of the surgeon on study.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for SMMS of cutaneous melanoma (stage 0 through stage IIc per American Joint Committee on Cancer [AJCC] criteria)
* Age >= 18 years at time of consent
* Initial tumor biopsy is PRAME positive or PRAME testing was not done. PRAME testing must be planned if not done
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Initial biopsy was PRAME negative
* Incarcerated persons
* Patient with severe, active co-morbidity that would preclude a SMMS of cutaneous melanoma (stage 0 through stage IIc per AJCC criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Margin status | During slow Mohs micrographic surgery (SMMS) procedure
  Margin status (positive, negative, or uncertain) will be evaluated from hematoxylin and eosin (H&E)/SOX-10 + preferentially expressed antigen in melanoma (PRAME) stained sections versus H&E/SOX-10 stained sections. For PRAME stained sections, margins will be considered positive when > 75% PRAME+ malignant cells at the tissue margin are observed. The McNemar's test will be used to compare the margin status between the predetermined gold-standard (i.e., H&E/SOX-10) and H&E/SOX-10 + PRAME.

SECONDARY OUTCOMES:
Presence of PRAME+ suprabasilar melanocytes in the tissue sections | During SMMS procedure
  Will be reported using descriptive statistics, including frequency tables as appropriate.
Density of PRAME+ cells | During SMMS procedure
  Will be reported as a quartile system (0% positive, 1-25% positive, 26-50% positive, 51-75% positive and > 75% positive). Will be reported using descriptive statistics, including frequency tables as appropriate.
Number of stages needed for clear margins | During SMMS procedure
  Will be reported using descriptive statistics, including frequency tables as appropriate.
Local recurrence of the excised melanoma | Up to 5 years following SMMS
  Will be reported using descriptive statistics, including frequency tables as appropriate.
Incidence of regional and distant metastases | Up to 5 years following SMMS
  Will be reported using descriptive statistics, including frequency tables as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Eisen, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States